CLINICAL TRIAL: NCT06218407
Title: Development and Evaluation of Computerized Chemosensory Based Orbitofrontal Networks Training for Treatment of Pain (CBOT-P)
Brief Title: Development and Evaluation of Computerized Chemosensory Based Orbitofrontal Networks Training for Treatment of Pain
Acronym: CBOT-Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evon Medics LLC (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Howard University (Other); Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CBOTNS125745; 1R44NS125745-01A1 (NIH)
Record Dates: First submitted 2024-01-08; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain; Low Back Pain
Keywords: Chronic Pain (CP); Pain; Negative Affect (NA); Cognitive Impairments; Attenuation of Structural Brain loss in CP with high NA; PACS outcome; Orbitofrontal cortex; Chemosensory-Based Orbitofrontal Networks Training
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Pain; Cognitive Dysfunction | interventions — caryophyllene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) short-burst paradigm (Experimental): CBOT consists of repetitive cycles of olfactory stimulation and tasks daily for 14 days.
  Interventions: Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) short burst paradigm
- Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) long-burst paradigm (Experimental): CBOT consists of repetitive cycles of olfactory stimulation and tasks daily for 14 days.
  Interventions: Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) long burst paradigm
- CBOT plus (CBOT + beta caryophyllene [BCP]) (Experimental): CBOT device enhanced with BCP
  Interventions: Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training plus beta caryophyllene (CBOT-Plus)
- Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) (Sham Comparator): CBOT device without BCP enhancement as control for BCP
  Interventions: Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT)

INTERVENTIONS:
Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) short burst paradigm — The CBOT device is designed to stimulate intensive neural activity in the medial orbitofrontal regions over long periods of time.
  Other Names: CBOT-Short
  Arms: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) short-burst paradigm
Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) long burst paradigm — The CBOT device is designed to stimulate intensive neural activity in the lateral orbitofrontal regions and networks over long periods of time.
  Other Names: CBOT-Long
  Arms: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) long-burst paradigm
Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training plus beta caryophyllene (CBOT-Plus) — CBOT device enhanced with BCP.
  Other Names: CBOT Plus
  Arms: CBOT plus (CBOT + beta caryophyllene [BCP])
Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) — CBOT device administering continuous olfactory stimuli (i.e., not programmed for short or long burst), and without BCP enhancement.
  Other Names: CBOT
  Arms: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT)

SUMMARY:
The overarching goal of this study phase, Phase I component is to configure Computerized Chemosensory-Based Orbitofrontal Networks Training (CBOT) into Computerized Chemosensory-Based Orbitofrontal Networks Training for Treatment of Pain CBOT-Pain (or CBOT-P) for rapid and sustained reduction of Pain, Negative Affect (NA) and Cognitive Impairments. The investigators aimed at first establishing if stimulation parameters targeting key olfactory regions, and their associated networks, paired with tasks that synergistically activate the orbitofrontal cortex (OFC) would have significantly different acute (< 7 days) effects in pain and NA intensity reductions. The hypothesis is that the short burst paradigm will more effectively activate the medial OFC and its functional connectivity with medial temporal affective networks, and result in greater reduction of affect and pain severity ratings after 7 days. The investigators will further examine if enhancing the odor regimen with beta-caryophyllene (BCP) content would have more dramatic effects in acute relief of pain, NA, and cognition.

Aim 1.1: To optimize CBOT-P stimulation parameters and olfactory stimulants for pain, affect and cognition in CP with and without high NA. This is a 14-day prospective study, in which fMRI and rs-fMRI will be acquired at baseline and day 7 during exposure to short vs long-burst CBOT stimulations. This is followed by daily treatment with short-burst versus long-burst CBOT paradigm over 14 days, during which pain and NA measures will be recorded daily by the subjects, and assessed by train research staff at baseline, day 7 and day 14.

Aim 1.2: To determine if CBOT regimen optimized with BCP content produces stronger and faster pain and affective response. This is a 14-day prospective study design, in which daily treatment of CBOT-PLUS (i.e., CBOT with BCP) will be compared against daily treatment with CBOT without BCP enhancement (CBOT). Subjects and clinicians are blinded to the assigned arms. Pain and NA measures will be recorded daily by the subjects and assessed by trained research staff at baseline and day 14.

DETAILED DESCRIPTION:
The Development and Evaluation of Computerized Chemosensory-Based Orbitofrontal Networks Training for Treatment of Pain (CBOT-P) is a project to develop an effective, scalable, user-friendly, and homebased neuromodulatory platform for broad-spectrum treatment of chronic pain conditions with associated negative affect and cognitive impairments.

The small business, Evon Medics created the olfactory pulsing technology called Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT-P) to enable home-based modulation of the OFC and subcortical limbic structures for treatment of pain and negative affect. In a stakeholder value canvassing exercise CP sufferers and pain doctors unanimously desire new non-invasive, home-based, safe, and effective interventions that can reduce pain severity by more than 10%, suggesting that current treatments have limitations. Anterograde and retrograde anatomical tracings have been used to demonstrate direct (monosynaptic) anatomical connection between the OFC and the descending inhibitory pain nodes at the midbrain periaqueductal gray matter (PAG). Transition to CP is marked by weakened modulation of the PAG-descending inhibition.

In this study phase, Phase I of this Fast-Track SBIR application, the investigators will (a) configure CBOT-P regimen and stimulation parameters for faster onset of mood elevating and analgesic effects, focusing on Chronic Low Back Pain populations and (b) establish its neural mechanism of action through target-engagement studies of OFC activity and functional connectivity with other pain regulating regions at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-85.
2. Pain duration > 6 months.
3. Must meet the minimum criteria for cognitive function using the PROMIS 2-item cognitive screener >3.
4. Average pain score of > 5/10, with low back pain being the primary pain site.
5. CLBP (chronic low back pain) meeting Quebec Task Force Classification System Categories I-III.
6. Evidence of a prior lumbar spine X-ray to rule out red flags, such as infection, tumor, or fracture.
7. For those taking opioids (the opioid subgroup), participants must be prescribed opioids currently for at least 3 consecutive months prior to enrollment. Such patients must be on opioids for a minimum of three months, taking them daily or intermittently during the week.
8. Subject must agree that opioids cannot be increased during the study.
9. No substance use disorder (SUD), except tobacco, in the past year based on substance screening surveys and frequent urine toxicology screens.
10. No acute suicidality, mania, or psychosis. This will be assessed at study entry which will also include a review of history in the EHR, Structured Clinical Interview for Psychiatric Disorders (SCID-5) and Columbia Suicide Severity Rating Scale (C-SSRS) and -
11. Participants must sign IRB-approved consent.

Exclusion Criteria:

1. Back surgery within the past six months.
2. Active worker's compensation or litigation claims.
3. New pain and/or psychiatric treatments within 2 weeks of enrollment.
4. Intent to add new or increase pain treatments during the study period, such as back surgery, nerve block procedures, or medications.
5. Intent to add new psychiatric treatments during the first 3 months of the study.
6. Any clinically unstable systemic illness that is judged to interfere with the trial.
7. History of cardiac, nervous system, or respiratory disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for respiratory depression.
8. Non-ambulatory status.
9. Pregnancy or the intent to become pregnant during the study. Women of childbearing age will have urine pregnancy testing at enrollment and monthly.
10. Anosmia or significant nasal disease
11. Contraindications to MRI
12. Stroke or TBI (traumatic brain injury).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Relative changes in blood oxygen level dependent (BOLD) signals from fMRI of orbitofrontal brain regions in response to short durations (i.e., short-bursts) and to long durations (i.e., long-bursts) of repetitive odor stimulations. Aim 1.1 | Baseline
  The blood-oxygen-level-dependent (BOLD) signal, acquired in functional Magnetic Resonance Imaging (fMRI), is a reflection of changes in deoxyhemoglobin driven by localized changes in brain blood flow and blood oxygenation, which are coupled to underlying neuronal activity by a process termed neurovascular coupling. In the context of pain disorders, fMRI has been used to study changes in brain function related to pain and to responses to interventions for pain. In the context of this study, positive BOLD signals in the brain region of interest, seen in response to odorant stimuli, represent a decrease in deoxyhemoglobin and thus an over-oxygenation of the responding region. Studies have shown that these changes in BOLD signals correlate with brain activity - with positive increase in BOLD signal reflective of increased brain activity and decreased BOLD signal reflective of reduced brain activity.
Changes in the resting-state functional connectivity between midbrain and corticolimbic brain regions Aim 1.1 | Baseline to day 7
  Changes in the resting-state functional connectivity between midbrain and corticolimbic brain regions, defined as correlations between low-frequency oscillations in the functional magnetic resonance (fMRI) blood oxygenation level dependent signal in these brain regions of interest acquired in the absence of a cognitive task. As a correlation, this measure ranges from -1 to 1. The higher the value (above zero) between two brain regions the more positively correlated are their low-frequency oscillations of fMRI blood oxygenation level dependent signals. The lower their value (below zero) between brain regions the more negatively correlated are their low-frequency oscillations of fMRI blood oxygenation level dependent signals.
Patient Reported Outcomes Measurement Information System (PROMIS) Numeric Rating Scale v1.0 - Pain Intensity Aim 1.1 | Baseline to day 7
  Change in 11-point score PROMIS Numeric Rating Scale v1.0 - Pain Intensity from baseline.
  The Numeric Rating Scale measures each consist of a single item rating pain on average over the past 7 days from 0 (no pain) to 10 (worst pain).
Positive and Negative Affect Schedule (PANAS) rating scale Aim 1.1 | Baseline to day 7
  Change in negative affect score from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Relative changes in blood oxygen level dependent (BOLD) signals from fMRI of orbitofrontal brain regions in response to short durations (i.e., short-bursts) and to long durations (i.e., long-bursts) of repetitive odor stimulations. Aim 1.1 | 7 days after baseline
  The blood-oxygen-level-dependent (BOLD) signal, acquired in fMRI, is a reflection of changes in deoxyhemoglobin driven by localized changes in brain blood flow and blood oxygenation, which are coupled to underlying neuronal activity by a process termed neurovascular coupling. In the context of pain disorders, fMRI has been used to study changes in brain function related to pain and to responses to interventions for pain. In the context of this study, positive BOLD signals in the brain region of interest, seen in response to odorant stimuli, represent a decrease in deoxyhemoglobin and thus an over-oxygenation of the responding region. Studies have shown that these changes in BOLD signals correlate with brain activity - with positive increase in BOLD signal reflective of increased brain activity and decreased BOLD signal reflective of reduced brain activity.
Patient Reported Outcomes Measurement Information System (PROMIS) Numeric Rating Scale v1.0 - Pain Intensity Aim 1.2 | Baseline to day 7
  Change in 11-point score PROMIS Numeric Rating Scale v1.0 - Pain Intensity from baseline.
  The Numeric Rating Scale measures each consist of a single item rating pain on average over the past 7 days from 0 (no pain) to 10 (worst pain).
Positive and Negative Affect Schedule (PANAS) rating scale Aim 1.2 | Baseline to day 7
  Change in negative affect score from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Patient Reported Outcomes Measurement Information System (PROMIS) Numeric Rating Scale v1.0 - Pain Intensity Aim 1.1 | Baseline to day 14
  Change in 11-point score PROMIS Numeric Rating Scale v1.0 - Pain Intensity from baseline.
  The Numeric Rating Scale measures each consist of a single item rating pain on average over the past 7 days from 0 (no pain) to 10 (worst pain).
Positive and Negative Affect Schedule (PANAS) rating scale Aim 1.1 | Baseline to day 14
  Change in negative affect score from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Changes in the resting-state functional connectivity between midbrain and corticolimbic brain regions Aim 1.1 | Baseline to 14
  Changes in the resting-state functional connectivity between midbrain and corticolimbic brain regions, defined as correlations between low-frequency oscillations in the functional magnetic resonance (fMRI) blood oxygenation level dependent signal in these brain regions of interest acquired in the absence of a cognitive task. As a correlation, this measure ranges from -1 to 1. The higher the value (above zero) between two brain regions the more positively correlated are their low-frequency oscillations of fMRI blood oxygenation level dependent signals. The lower their value (below zero) between brain regions the more negatively correlated are their low-frequency oscillations of fMRI blood oxygenation level dependent signals.
Patient Reported Outcomes Measurement Information System (PROMIS) Numeric Rating Scale v1.0 - Pain Intensity Aim 1.2 | Baseline to day 14
  Change in 11-point score PROMIS Numeric Rating Scale v1.0 - Pain Intensity from baseline.
  The Numeric Rating Scale measures each consist of a single item rating pain on average over the past 7 days from 0 (no pain) to 10 (worst pain).
Positive and Negative Affect Schedule (PANAS) rating scale Aim 1.2 | Baseline to day 14
  Change in negative affect score from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.1 - Pain Interference scores. Aim 1.1 | Baseline to day 7
  Change in PROMIS Short Form v1.1 - Pain Interference scores.
  The PROMIS Pain Interference Short Form 4a is consists of 4 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 4; the highest possible raw score is 20.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Anxiety scores Aim 1.1 | Baseline to day 7
  Change in PROMIS Short Form v1.0 - Anxiety scores
  The PROMIS Anxiety 1a is consists of 55 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 55; the highest possible raw score is 275.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Sleep Disturbance scores Aim 1.1 | Baseline to day 7
  Change in PROMIS Short Form v1.0 - Sleep Disturbance scores
  The PROMIS Sleep Disturbance v1.0 is consists of 26 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 26; the highest possible raw score is 130.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Pittsburgh Sleep Quality Index (PSQI) Aim 1.1 | Baseline to day 7
  Change in Pittsburgh Sleep Quality Index (PSQI) scores
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. Each component generates a score from 0-3 where higher scores indicate poorer sleep outcomes.
  In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
  A global score above 5 indicates poor sleep quality.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Anxiety scores Aim 1.2 | Baseline to day 7
  Change in PROMIS Short Form v1.0 - Anxiety scores
  The PROMIS Anxiety 1a is consists of 55 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 55; the highest possible raw score is 275.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Sleep Disturbance scores Aim 1.2 | Baseline to day 7
  Change in PROMIS Short Form v1.0 - Sleep Disturbance scores
  The PROMIS Sleep Disturbance v1.0 is consists of 26 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 26; the highest possible raw score is 130.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Pittsburgh Sleep Quality Index (PSQI) Aim 1.2 | Baseline to day 7
  Change in Pittsburgh Sleep Quality Index (PSQI) scores
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. Each component generates a score from 0-3 where higher scores indicate poorer sleep outcomes.
  In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
  A global score above 5 indicates poor sleep quality.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v2.0 - Physical Function Aim 1.2 | Baseline to day 7
  Change in PROMIS Short Form v2.0 - Physical Function score
  PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. The PROMIS short form v2.0 Physical function instrument is consists of 22 questions, each question has five response options ranging in value from one to five. The lowest possible raw score is 22 and the highest possible raw score is 113.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Global Impression of Change Aim 1.2 | Baseline to day 7
  Change in Patient Global Impression of Change score
  The Patient Global Impression of Change scale is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time. It is a patient-reported outcome measure that can be used to assess treatment benefit in clinical trials or practice. It is based on the Clinical Global Impression of Change scale, which is an observer-rated scale of symptom severity and treatment response. The scale ranges from 1 (no change or worse) to 7 (a great deal better).
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.1 - Pain Interference scores. Aim 1.1 | Baseline to day 14
  Change in PROMIS Short Form v1.1 - Pain Interference scores.
  The PROMIS Pain Interference Short Form 4a is consists of 4 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 4; the highest possible raw score is 20.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Anxiety scores Aim 1.1 | Baseline to day 14
  Change in PROMIS Short Form v1.0 - Anxiety scores
  The PROMIS Anxiety 1a is consists of 55 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 55; the highest possible raw score is 275.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Sleep Disturbance scores Aim 1.1 | Baseline to day 14
  Change in PROMIS Short Form v1.0 - Sleep Disturbance scores
  The PROMIS Sleep Disturbance v1.0 is consists of 26 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 26; the highest possible raw score is 130.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Pittsburgh Sleep Quality Index (PSQI) Aim 1.1 | Baseline to day 14
  Change in Pittsburgh Sleep Quality Index (PSQI) scores
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. Each component generates a score from 0-3 where higher scores indicate poorer sleep outcomes.
  In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
  A global score above 5 indicates poor sleep quality.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Anxiety scores Aim 1.2 | Baseline to day 14
  Change in PROMIS Short Form v1.0 - Anxiety scores
  The PROMIS Anxiety 1a is consists of 55 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 55; the highest possible raw score is 275.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Sleep Disturbance scores Aim 1.2 | Baseline to day 14
  Change in PROMIS Short Form v1.0 - Sleep Disturbance scores
  The PROMIS Sleep Disturbance v1.0 is consists of 26 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 26; the highest possible raw score is 130.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Pittsburgh Sleep Quality Index (PSQI) Aim 1.2 | Baseline to day 14
  Change in Pittsburgh Sleep Quality Index (PSQI) scores
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. Each component generates a score from 0-3 where higher scores indicate poorer sleep outcomes.
  In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
  A global score above 5 indicates poor sleep quality.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v2.0 - Physical Function Aim 1.2 | baseline to day 14
  Change in PROMIS Short Form v2.0 - Physical Function score
  PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. The PROMIS short form v2.0 Physical function instrument is consists of 22 questions, each question has five response options ranging in value from one to five. The lowest possible raw score is 22 and the highest possible raw score is 113.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Global Impression of Change Aim 1.2 | Baseline to day 14
  The Patient Global Impression of Change scale is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time. It is a patient-reported outcome measure that can be used to assess treatment benefit in clinical trials or practice. It is based on the Clinical Global Impression of Change scale, which is an observer-rated scale of symptom severity and treatment response. The scale ranges from 1 (no change or worse) to 7 (a great deal better).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Nwaokobia, Principal Investigator — Evon Medics LLC; Evaristus Nwulia, MD, Principal Investigator — Howard University; Tanya Alim, MD, Principal Investigator — Howar
Locations (1):
- Howard University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No